CLINICAL TRIAL: NCT04505527
Title: Variability of Movement on an Altered Inertial Dynamics Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0448-16-FB; P20GM109090 (NIH)
Record Dates: First submitted 2020-08-02; First posted 2020-08-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Older Adults; Fall Patients
Keywords: balance; gait; variability

STUDY DESIGN:
Intervention Model Description: Older adults will be screened and will be randomly assigned to three groups - (i) non-fallers, (ii) recurrent fallers - control group, and (iii) recurrent fallers - intervention group. A fourth group consisted of healthy young adults. This group will receive lateral stepping intervention and outcomes will be measured as a reference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Recurrent fallers - control group (Active Comparator): In this control arm, older adults will have a typical forward walking training that mirror the lateral stepping intervention: 3 days/week for 6 weeks, resulting in a total of eighteen sessions. Each session consists of six trials of 3 min forward walking. The participants can increase their pace at the start of each trial but may not decrease it at the next session.
  Interventions: Behavioral: Forward walking
- Recurrent fallers - intervention group (Experimental): In this experimental arm, older adults will have a lateral stepping intervention: 3 days/week for 6 weeks, resulting in a total of eighteen sessions. Each session consists of six trials of 3 min sideways walking across a 10 m walkway changing body direction at the ends, thus alternating lead and lag limbs. The participants can increase their pace at the start of each trial but may not decrease it at the next session.
  Interventions: Behavioral: Lateral stepping
- Older non-fallers intervention group (Experimental): In this experimental arm, older adults will have a lateral stepping intervention: 3 days/week for 6 weeks, resulting in a total of eighteen sessions. Each session consists of six trials of 3 min sideways walking across a 10 m walkway changing body direction at the ends, thus alternating lead and lag limbs. The participants can increase their pace at the start of each trial but may not decrease it at the next session.
  Interventions: Behavioral: Lateral stepping
- Younger adult control group (Active Comparator): Outcome measures from a young healthy group will also be measured as a reference. Will be used to compare outcome measured between older and young adults. Young adults will have a lateral stepping intervention: 3 days/week for 6 weeks, resulting in a total of eighteen sessions. Each session consists of six trials of 3 min sideways walking across a 10 m walkway changing body direction at the ends, thus alternating lead and lag limbs. The participants can increase their pace at the start of each trial but may not decrease it at the next session.
  Interventions: Behavioral: Lateral stepping

INTERVENTIONS:
Behavioral: Lateral stepping — Subjects will step laterally, changing direction every 10 m, thus alternating lead and lag limbs.
  Other Names: Sideways walking
  Arms: Older non-fallers intervention group; Recurrent fallers - intervention group; Younger adult control group
Behavioral: Forward walking — Subjects will have a typical forward walking
  Other Names: Typical walking
  Arms: Recurrent fallers - control group

SUMMARY:
The overall goal of this research is to compare the effects of two different exercise programs on gait function in older adults. The investigators want to determine if participation in lateral stepping exercise program for six weeks will improve gait functions compared to forward walking exercise program.

DETAILED DESCRIPTION:
The overall goal of this research is to compare the effects of two different exercise programs on gait function in older adults. It is expected that improved control of foot placement in the lateral stepping task will transfer to improved control during typical forward walking. Moreover, it is expected that lateral stepping gait training will have a greater effect on recurrent fallers older adults than on the non-fallers older adults and young adults. It is also expected that the above beneficial results will be retained in a follow-up test six weeks after completion of the intervention and will result in improvements in common clinical balance tests that are used to assess fall risk. Therefore, in the current proposal, older adults aged 65 years of age and over are being asked to participate.

ELIGIBILITY:
Inclusion Criteria:

Subjects must

* be aged between 19 and 35 for the young adult group
* be over 65 years of age for the older adult groups
* be independently residing in the community
* be able to provide informed consent
* be able to walk independently without an assistive device or 30 minutes in three-minute sections interspersed with rest periods.

The older participants must either have sustained two or more falls in the past year (i.e. Fallers) or not have sustained any falls in the past year (i.e. Non-Fallers).

Exclusion Criteria:

* Neurological disorder or progressive neurologic condition - epilepsy, Alzheimer disease and other dementias, stroke, multiple sclerosis, Parkinson's disease, brain infections, brain tumors.
* Movement disorder - ataxia, dystonia, Huntington's disease, myoclonus, Parkinson disease, progressive supranuclear palsy, Wilson disease.
* History of Cardiovascular events this includes any history of heart problems (such as heart attack, chest pain, or conditions which affect the heart's muscles, valves, or rhythm)
* Current injury or moderate to severe pain affecting the lower limbs, pelvis, back, trunk.
* Surgery within the past 6 months.
* Current participation in any other study that involves walking, balance, or training.

Medications will not prevent inclusion in the study however they will be recorded to enable consideration in subsequent post-hoc analyses.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Step width variability | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The standard deviation of step width. Step width was measured as the mediolateral distance between the locations of the sequential left and right heel strikes
Step length variability | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The standard deviation of step length. Step length was measured as the anteroposterior distance between the locations of the sequential left and right heel strikes.
Swing time variability | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The standard deviation of swing time. Swing time was measured as the time elapse during the swing phase of a leg.
Stride time variability | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The standard deviation of stride time. Stride time was measured as the time between 2 consecutive ipsilateral heel strikes.
Stance time variability | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The standard deviation of stance time. Stance time was measured as the time elapse during the stance phase of a leg.
Timed-Up-and-Go (TUG) | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The Timed-Up-and-Go test is used to assess mobility in older adults. It measures the time to get up from chair, walk 3 m, turn around, walk back, and sit down
Berg Balance Test (BBS) | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The Berg Balance Test (14 items, max score: 56) is used to measure the functional balance in older adults. It consists of 14 tasks performed in a standardized order with each task scored on a five-point scale according to quality or time ranging from "0" (lowest level of function) to "4" (highest level).

SECONDARY OUTCOMES:
Walking speed | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  Self-selected forward walking and sideways walking speed
Falls Efficacy Scale-International (FES-I) | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The Falls Efficacy Scale-International (FES-I) questionnaire (16 items, max score: 64) is used to assess confidence in the performance of activities relevant to daily life. Participants rate 16 individual activities on a scale from 1 (not at all concerned) to 4 (very concerned).

OTHER OUTCOMES:
Brief Pain Inventory - short form (BPI) | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The short form of Brief Pain Inventory score (BPI) (4 Pain severity items, max score: 40; 7 Pain interference items, max score: 70) is used to measure the impact of pain on daily functions. Higher score suggests higher pain intensity (severity), and/or higher impact of pain on functioning (interference).
Mini-Mental State Examination (MMSE) | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The Mini-Mental State Examination (MMSE) (11 items, max score: 30) is used to measure cognitive impairment. It consists of 11 questions grouped into 7 cognitive tasks. A score of 30 suggests no presence of cognitive impairment.
Geriatric Depression Scale - short form (GDS) | Baseline and Post-Intervention: immediate, and 6 weeks after the completion of the intervention
  The Geriatric Depression Scale - short form (GDS) (15 items, max score: 15) is used to measure self-rated depressive symptoms of depression. A score of 5 or more suggests depression.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Skiadopoulos, PhD, Principal Investigator — Research Associate; Nicholas Stergiou, PhD, Study Director — Assistant Dean
Locations (1):
- University of Nebraska-Omaha, Biomechanics Research Building, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Skiadopoulos A, Stergiou N. Risk-of-falling related outcomes improved in community-dwelling older adults after a 6-week sideways walking intervention: a feasibility and pilot study. BMC Geriatr. 2021 Jan 14;21(1):60. doi: 10.1186/s12877-021-02010-6. PMID 33446112